CLINICAL TRIAL: NCT05888077
Title: Extracorporeal Shock Wave Lithotripsy Using Latest Lithotripter and Laser Lithotripsy for Difficult Bile Duct Stones
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Other Study IDs: ESWL_LL
Record Dates: First submitted 2023-05-25; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Bile Duct Stenosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

INTERVENTIONS:
Other: ESWL_LL — Extracorporeal shock wave lithotripsy using latest lithotripter and laser lithotripsy for difficult Bile duct stones

SUMMARY:
When conventional endoscopic treatment of bile duct stones is impossible or fails, advanced endoscopy assisted lithotripsy can be performed by electrohydraulic lithotripsy (EHL), laser lithotripsy, or extracorporeal shock wave lithotripsy (ESWL). No systematic review has compared efficacy and safety between these techniques.

DETAILED DESCRIPTION:
Extracorporeal shock wave lithotripsy (ESWL) and Laser Lithotripsy (LL) have emerged as alternate treatment options for difficult common bile duct (CBD) stones. There is limited data on efficacy and safety of the latest Dornier delta III lithotripter. This study examined the efficacy of ESWL by Dornier delta III & Laser lithotripsy in terms of stone clearance rate, number of sessions required and safety in a large cohort of patients.

The initial lithotripter models used electrohydraulic energy and required general anesthesia, prone positioning, and water immersion. High clearance rates were reported, but newer models were then developed with use of electromagnetic coils, better focussing, use of a water cushion instead of water immersion, use of ultrasound and then later of digitalised X ray for localisation. The ductal clearance of ESWL is upto 90%. Known complications of this procedure are cholangitis and pancreatitis which occur at the rate of 9-14% apart from minor adverse effects such as pain and local hematoma formation. In a single randomised study that compared intracorporeal lithotripsy(ILL) versus extracorporeal lithotripsy, ILL was found more effective than ESWL in terms of stone clearance rate and treatment duration. However, the lithotripters used in the previous studies were of previous generations, and also commonly used for kidney stones as well. The current study is the first to use the Dornier delta III for the same.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stones that could not be extracted by conventional methods such as biliary sphincterotomy, balloon, basket or mechanical lithotripsy.
* Patients with biliary stones larger than 15mm.
* Intrahepatic or cystic duct stones.

Exclusion Criteria:

* Pregnancy.
* Coagulopathy which cannot be corrected.
* Ongoing cholangitis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study is a retrospective analysis of prospectively collected data from the Asian Institute of gastroenterology, India, between January 2019 to December 2022. All patients undergoing biliary ESWL and LL from January 2019 to December 2022 were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy ESWL and Laser lithotripsy | One year
  Efficacy of ESWL by Dornier delta III & Laser lithotripsy in terms of stone clearance rate

IPD SHARING:
Plan to Share IPD: No